CLINICAL TRIAL: NCT05605990
Title: Clinical Application and Validation of Innovative Tourniquet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Chou-Ching Lin, Professor, National Cheng-Kung University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB No.A-BR-111-011
Record Dates: First submitted 2022-10-25; First posted 2022-11-04 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Compartment Syndrome of Forearm

STUDY DESIGN:
Intervention Model Description: We will recruit 160 nurses in high-risk units of the hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nurse group (Experimental): Using an innovative tourniquet (Acusense Nonpneumatic tourniquet) for the standard of care
  Interventions: Device: Innovative tourniquet (Acusense Nonpneumatic tourniquet)

INTERVENTIONS:
Device: Innovative tourniquet (Acusense Nonpneumatic tourniquet) — To use this innovative tourniquet before collecting blood samples, and setting IV catheter. We also use this innovative tourniquet to occlude the flow of blood.

SUMMARY:
Background: Tourniquets are the basic equipment for nurses to perform blood draws, and venous indwelling needles for congestion, or for hemostasis. Therefore, forgetting to remove the tourniquet is a common problem that leads to blood circulation being blocked, and even severe tissue necrosis occurred.

Purpose: The study aimed to evaluate whether this innovative tourniquet could prevent forgetting to remove the tourniquet, and improve the satisfaction of care.

Research design: This clinical research trial was a quasi-experimental study designed for a single group with pre-and post-test. We will recruit 160 nurses in high-risk units of the hospital. The delay in removing the tourniquet as our study outcome is defined as the removing time delay of one minute.

Expected results: The research results will provide some evidence of the efficacy of intelligent tourniquets.

ELIGIBILITY:
Inclusion Criteria: Nurse group: We included nurses who have working experience of more than 3 months, and are willing to use an innovative tourniquet.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Preventing the forgetting to remove the tourniquet | A three months period
  Forgetting to remove the tourniquet is defined as the optimal removing time to delay of one minute.
Enhancing nurses' satisfaction | A three months period
  The Likert Scale asks how much a person agrees or disagrees with a particular statement or question. It is usually made up of a 5-point rating scale ranging from 1 and 5 with 10-item.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng Kung University Hospital, College of Medicine, National Cheng Kung University, Tainan, Taiwan, Tainan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Gorski LA, Hadaway L, Hagle ME, Broadhurst D, Clare S, Kleidon T, Meyer BM, Nickel B, Rowley S, Sharpe E, Alexander M. Infusion Therapy Standards of Practice, 8th Edition. J Infus Nurs. 2021 Jan-Feb 01;44(1S Suppl 1):S1-S224. doi: 10.1097/NAN.0000000000000396. No abstract available. PMID 33394637
- [Result] Lee C, Porter KM, Hodgetts TJ. Tourniquet use in the civilian prehospital setting. Emerg Med J. 2007 Aug;24(8):584-7. doi: 10.1136/emj.2007.046359. PMID 17652690
- [Result] Pinkerton C. New technology enhances expertise of vascular access team. Can Nurse. 2009 Feb;105(2):21-2. No abstract available. PMID 19263937
- [Result] Duignan KM, Lamb LC, DiFiori MM, Quinlavin J, Feeney JM. Tourniquet use in the prehospital setting: Are they being used appropriately? Am J Disaster Med. 2018;13(1):37-43. doi: 10.5055/ajdm.2018.0286. PMID 29799611